CLINICAL TRIAL: NCT01371084
Title: Pilot Study to Test the Efficacy of a Worksite Intervention for Reducing Daily Sedentary Time and Improving Risk Factors for Cardiometabolic Disease Among Sedentary, Overweight, Full-time Working Adults
Brief Title: Pedal@Work: A Worksite Wellness Program
Acronym: Pedal@Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Lucas J. Carr, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 212112
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity treatment group (Experimental): Participants randomized to the intervention group will be provided access to a portable pedal exercise machine, a pedometer and a worksite wellness motivational website for 12 weeks. As part of this website, participants will be emailed behavioral intervention materials a maximum of three times per week targeted at reducing sedentary time.
  Interventions: Behavioral: Pedal@Work
- Wait List Control (Placebo Comparator)
  Interventions: Behavioral: Pedal@Work Worksite Wellness

INTERVENTIONS:
Behavioral: Pedal@Work Worksite Wellness — Participants randomized to the intervention group will be provided access to a portable pedal exercise machine, a pedometer and a worksite wellness motivational website for 12 weeks. As part of this website, participants will be emailed behavioral intervention materials a maximum of three times per week targeted at reducing sedentary time.
  Arms: Wait List Control
Behavioral: Pedal@Work — Worksite wellness program.
  Arms: Physical activity treatment group

SUMMARY:
The primary aim of this pilot study is to test the efficacy of a worksite intervention for reducing daily sedentary time and improving risk factors for cardiometabolic disease (e.g., measures of adiposity, anthropometrics, cardiorespiratory fitness) among sedentary, overweight, full-time working adults as compared to a waitlist control. A secondary aim will be to test pedal time at work as a measure of compliance with the intervention.

DETAILED DESCRIPTION:
Recent research indicates prolonged sedentary behaviors such as computer use and workplace sitting are particularly damaging resulting in increased risk for chronic diseases such as cardiovascular disease, type 2 diabetes and obesity. Few interventions have been tested with the specific purpose of reducing sedentary time to improve risk factors for cardiometabolic diseases. The primary aim of this pilot study is to test the efficacy of a worksite intervention for reducing daily sedentary time and improving risk factors for cardiometabolic disease (e.g., measures of adiposity, anthropometrics, cardiorespiratory fitness) among sedentary, overweight, full-time working adults as compared to a waitlist control. A secondary aim will be to test pedal time at work as a measure of compliance with the intervention. Participants will be followed for 12 weeks and randomized to either a treatment or wait list control group which will have the option to crossover into the intervention after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 21 and 65 years
* Sedentary (engaging in moderate intensity physical activity for less than 60 minutes per week)
* Working full time (35+ hours/week) at a sedentary desk dependant occupation
* Overweight (Body Mass Index > 25.0 kg/m2 but less than 40.0 kg/2)
* Apparently healthy as assessed by a health history screening survey
* Devoid of overt complicated or acute cardiovascular, metabolic, respiratory, or neurological diseases
* Free from exercise/physical activity limitations

Exclusion Criteria:

* Adults with significant health problems exacerbated by exercise, such as uncontrolled hypertension, diabetes, orthopedic limitations, etc. will be excluded from the study. Note, with physician approval and adequate control of these health problems, these conditions will not necessarily preclude participation.
* Being unable to exercise

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Step Watch - Physical Activity Minutes | 12 weeks between baseline and post-intervention follow up
  Participants will wear a Step Watch monitor for 7 days at baseline and post-intervention. The intervention time period is 12 weeks.

SECONDARY OUTCOMES:
Cardiometabolic Risk | 12 weeks between baseline and post-intervention follow up
  Cardiometabolic risk will be assessed by blood pressure, heart rate, cardiopulmonary fitness, lipids, waist circumference, BMI, and percent body fat

CONTACTS AND LOCATIONS:
Overall Officials: Lucas J Carr, Ph.D., Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

REFERENCES:
- [Derived] Carr LJ, Karvinen K, Peavler M, Smith R, Cangelosi K. Multicomponent intervention to reduce daily sedentary time: a randomised controlled trial. BMJ Open. 2013 Oct 18;3(10):e003261. doi: 10.1136/bmjopen-2013-003261. PMID 24141969